CLINICAL TRIAL: NCT06103565
Title: Electronic Health Record Nudges to Improve Quality of Care in Heart Failure
Brief Title: EHR Nudges to Improve Quality of Care in HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Faraz Ahmad, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00214805
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Heart Failure, Systolic; Quality of Health Care; Pharmacists; Medication Adherence
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active clinical decision support tool for pharmacists (Other): In this single arm, pilot feasibility study, pharmacists with be exposed to a clinical decision support tool to facilitate monitoring adherence to GDMT for patients with heart failure with reduced ejection fraction
  Interventions: Other: Clinical Decision Support Tool

INTERVENTIONS:
Other: Clinical Decision Support Tool — Clinical decision support tool to enable pharmacists to monitor adherence to guideline-directed medical therapy for patients with heart failure with reduced ejection fraction

SUMMARY:
The purpose of this pilot feasibility study is to test a pharmacist-facing clinical decision support tool designed to increase adherence to guideline-directed medical therapy and evaluate the tool using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) evaluation framework.

DETAILED DESCRIPTION:
Heart failure (HF) is a common, morbid, and costly condition with an enormous toll on health and the health care system in the US. Unlike other HF types, for patients with HFrEF decades of high quality, randomized controlled trials have demonstrated numerous interventions-including medications, devices, and cardiac rehabilitation-that improve quality of life, lengthen survival, and reduce hospitalizations. Despite the substantial evidence, many patients with HFrEF do not receive optimal guideline-directed medical therapy (GDMT) as shown by several US quality registries dating back to 2009. Contributors to gaps in care quality have been shown to include patient-level (i.e., illness severity, race/ethnicity, socio-economic status), clinician-level (i.e., lack of knowledge, clinical inertia), and health system-level (i.e., lack of care coordination) factors.

Pharmacist-led clinics in several health systems and studies have been shown to lead to high rates of GDMT intensification. This finding is consistent with decades of research in HF and other conditions in which more resources allocated to disease management can improve quality of care. Yet, little data exist on adherence to optimal GDMT after completion of an intensive disease management program.

Northwestern Medicine is a large, integrated system that operates multiple pharmacist-led clinics to optimize GDMT in patients with HFrEF. Once patients reach the maximum level of intensification, they complete the program and are no longer actively followed by the pharmacist team. The adoption of electronic health records (EHRs) and integration of novel data sources, such as prescription fill data from third-party vendors, create the opportunity to implement strategies to monitor adherence over time and intervene when adherence declines. Clinical decision support nudges in the EHR are inexpensive strategies that have been shown in clinical areas outside of HF to increase adherence to evidence-based therapies. Studies that use pharmacy fill data to monitor adherence to evidence-based care are rare given some of the technical challenges of accessing these data and using them for clinical decision support tools.

In this pilot feasibility study, we aim to develop and test a pharmacist-facing clinical decision support tool designed to increase adherence to GDMT and evaluate the tool using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) evaluation framework.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacist at Northwestern Medicine participating in the Medication Adjusted to Target (MAT) Clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Reach | 2-months
  Percentage of alerts in which the pharmacist contacts the patient to discuss the low medication adherence rate

SECONDARY OUTCOMES:
Adoption | 2-months
  Percentage of pharmacists who contact at least 50% of eligible patients
Implementation | After the end of the 2-month intervention period
  Qualitative interviews will be conducted to evaluate acceptability, appropiateness, and feasibility

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small number of participants and the inability to fully de-identify the data, IPD will only be share with researchers with an appropriate data use agreement in place.